CLINICAL TRIAL: NCT04772157
Title: Evaluation of the Siemens POC HS CTn-I Test System
Brief Title: Safe Emergency Department DIscharGE Rate (SEIGE)
Acronym: SEIGE
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Siemens Healthineers (Unknown)
Responsible Party: Sponsor
Other Study IDs: SEIGE
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Myocardial Infarction; Acute Coronary Syndrome
Keywords: Troponin; acute myocardial injury; acute myocardial infarction; Siemens POC; Siemens POC Atellica® VTLi; Siemens POC HS cTn-I
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma tested on the Siemens POC HS cTn-I Analyzer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort: Study population: Prospective, observational cohort study of consecutives patients (goal, 1000 patients over 4 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin Healthcare / Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
  Interventions: Diagnostic Test: Cardiac Troponin Testing

INTERVENTIONS:
Diagnostic Test: Cardiac Troponin Testing — Lithium heparin whole blood and plasma samples will be measured with Siemens POC High Sensitivity Troponin-I Test System.

SUMMARY:
The Siemens POC High Sensitivity Troponin-I Test System is an in vitro diagnostic test for the quantitative measurement of cardiac troponin I (cTn-I) in fresh human capillary (fingerstick) whole blood, and lithium-heparinized venous whole blood or plasma, to be used by healthcare professionals at the point of care (POC) as well as in the clinical laboratory.

The Siemens POC High Sensitivity Troponin-I Test System is to be used as an aid in the diagnosis of myocardial infarction (MI).

DETAILED DESCRIPTION:
Study purpose/objective:

* Evaluate the clinical performance of the Siemens POC HS cTn-I test system for the diagnosis and rule out of AMI in patients presenting to the emergency department in whom serial cTnI measurements are obtained on clinical indication.
* Correlate the blood and plasma outcomes on the Siemens POC HS cTn-I test system as function of the corresponding hematocrit (Hct) values.

Hypothesis: The Siemens POC HS cTn-I Test System will offer an excellent diagnostic performance for acute myocardial injury and acute myocardial infarction, as well as expedite the risk stratification of patients for early discharge from the emergency department.

ELIGIBILITY:
Inclusion Criteria:

1. Presents to the ED, or ambulatory care center equivalent, with signs or symptoms suspicious of a possible ACS event.
2. Baseline cTn-I measurement and one additional cTn-I measurement at two hours after the first measurement.
3. At least one 12-lead electrocardiogram

Exclusion Criteria

1. Less than 21 years old
2. Pregnancy
3. Trauma
4. Declines to participate or has indicated that their blood/ medical information cannot be used for investigational purposes
5. Did not present through the ED
6. Transferred from an outside hospital or clinic.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients (goal, 1000 patients over 4 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin Healthcare / Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Examine the incidence of undetectable(<LoD), measurable (LoD - 99th percentile), and increased (>99th percentile) cTn concentrations for the Siemens POC HS cTn-I Test System | Day 1
  Examine the incidence of undetectable(<LoD), measurable (LoD - 99th percentile), and increased (>99th percentile) cTn concentrations for the Siemens POC HS cTn-I Test System in comparison to a high sensitivity cTnI assay (Abbott & Siemens Healthineers) to determine the potential impact on positivity rate, defined by sex-specific 99th percentiles.
Examine Concordance | Day 1
  Examine concordance (dis) between hs-cTnI in comparison to a high sensitivity (Abbott & Siemens Healthineers) cTnI assay
Examine the diagnostic performance for acute myocardial injury and acute myocardial infarction | Day 1
  Examine the diagnostic performance for a) acute myocardial injury and b) acute myocardial infarction based on various diagnostic strategies using hs-cTnI measurement(s), as follows:
  1. Single measurement strategies
     1. Limit of detection (LoD)
     2. Concentration threshold tailored to meet a clinical need: Derive an optimal rule-out ng/L cutoff for Siemens POC HS cTn-I Test System.
  2. Accelerated serial sampling (0/2h protocol)
     1. Using the both sex-specific and overall 99th percentiles
     2. Delta (absolute concentration serial change value, 0-2h) analysis
Describe the incidence, clinical characteristics and outcomes of patients with and without hs-cTnI increases above the sex-specific 99th percentile URLs | Day 1
  Describe the incidence, clinical characteristics and outcomes of patients with and without hs-cTnI increases above the sex-specific 99th percentile URLs, including patients categorized with acute myocardial injury and acute myocardial infarction, including type 1 and 2 myocardial infarction following the 4th Universal Definition of Myocardial Infarction.
Impact on the incidence of myocardial injury and myocardial infarction diagnoses. | Day 1
  Examine the potential impact on the incidence of myocardial injury and myocardial infarction diagnoses using hs-cTnI upon clinical practice implementation with a comparison to the hospital's final ICD-10 code diagnosis of type 1 and type 2 MIs.

SECONDARY OUTCOMES:
All-cause mortality | up to 30 days
  any death
Cardiac mortality | up to 30 days
  death due to cardiac reasons
Adjudicated index acute myocardial infarction according to 4th UDMI | on admission
  acute myocardial infarction, including sub-types following the Fourth Universal Definition of Myocardial Infarction
Safety Outcome - MACE | 30 days
  Major Adverse Cardiovascular Event - cardiac death, myocardial infarction, revascularization, congestive heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Fred S Apple, PhD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare Research Institute / Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096
- [Derived] Apple FS, Smith SW, Greenslade JH, Sandoval Y, Parsonage W, Ranasinghe I, Gaikwad N, Schulz K, Stephensen L, Schmidt CW, Okeson B, Cullen L; SAMIE Investigators. Single High-Sensitivity Point-of-Care Whole-Blood Cardiac Troponin I Measurement to Rule Out Acute Myocardial Infarction at Low Risk. Circulation. 2022 Dec 20;146(25):1918-1929. doi: 10.1161/CIRCULATIONAHA.122.061148. Epub 2022 Oct 31. PMID 36314160